CLINICAL TRIAL: NCT03080454
Title: The Effect of Treatment With the PathMaker Myoregulator Neuromodulation System Incorporating Trans-spinal Direct Current Stimulation (tsDCS) in Patients With Severe Hand Spasticity After Stroke
Brief Title: The Role of Trans-spinal Direct Current Stimulation (tsDCS) in Treating Patients With Hand Spasticity After Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: PathMaker Neurosystems Inc. (Industry); Dr. Zaghloul Ahmed (Unknown)
Responsible Party: Principal Investigator, Bruce Volpe, Principal Investigator, Northwell Health
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 15-110
Record Dates: First submitted 2017-03-06; First posted 2017-03-15 (Actual); Results first posted 2019-09-13 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2019-08

CONDITIONS: Stroke; Cerebrovascular Accident (CVA); Hemiparesis; Spasticity as Sequela of Stroke; Muscle Spasticity; Upper Extremity Paralysis
Keywords: stroke; CVA; Spasticity; hemiparesis; rehabilitation; trans-spinal direct current stimulation (tsDCS); non-invasive stimulation
MeSH Terms: conditions — Stroke; Paresis; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: All participants received both stimulation conditions (sham Doublestim and anodal Doublestim), separated by a 1-week washout period.
Who Masked: Participant
Masking Description: The sham stimulation condition preceded the anodal stimulation condition for all participants, and subjects were told they would receive both conditions, but were blinded to order of assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Doublestim (Placebo Comparator): Participants first received 5 daily, consecutive 20 min sessions of sham Doublestim (trans-spinal direct current stimulation + peripheral direct current stimulation). After a washout period of 1 week, they then received 5 daily, consecutive 20 min sessions of anodal Doublestim (trans-spinal direct current stimulation + peripheral direct current stimulation). For all participants, the sham condition preceded the anodal Doublestim condition.
  Interventions: Device: sham Doublestim
- Anodal Doublestim (Active Comparator): Participants first received 5 daily, consecutive 20 min sessions of sham Doublestim (trans-spinal direct current stimulation + peripheral direct current stimulation). After a washout period of 1 week, they then received 5 daily, consecutive 20 min sessions of anodal Doublestim (trans-spinal direct current stimulation + peripheral direct current stimulation). For all participants, the sham condition preceded the anodal Doublestim condition.
  Interventions: Device: anodal Doublestim

INTERVENTIONS:
Device: sham Doublestim — PathMaker MyoRegulator device
  Other Names: sham trans-spinal direct current stimulation + peripheral direct current stimulation (tsDCS + pDCS)
  Arms: Sham Doublestim
Device: anodal Doublestim — PathMaker MyoRegulator device
  Other Names: anodal trans-spinal direct current stimulation + peripheral direct current stimulation (tsDCS + pDCS)
  Arms: Anodal Doublestim

SUMMARY:
The purpose of this study is to evaluate if 5 consecutive sessions of PathMaker anodal DoubleStim treatment, which combines non-invasive stimulation of the spinal cord (tsDCS- trans-spinal direct current stimulation) and of the median nerve at the peripheral wrist (pDCS-- peripheral direct current stimulation), can significantly reduce spasticity of the wrist and hand after stroke.

ELIGIBILITY:
Inclusion Criteria:

1. First single focal unilateral hemisphere lesion with diagnosis verified by brain imaging (MRI or CT scans) that occurred at least 6 months prior
2. Cognitive function sufficient to understand the experiments and follow instructions
3. A Modified Ashworth Scale score between 1-3 points for wrist flexor and extensor muscles
4. A minimum of 15 degrees wrist passive range of motion (ROM) for wrist flexion and extension from wrist neutral position

Exclusion Criteria:

1. Focal brainstem or thalamic infarcts
2. Prior surgical treatments for spasticity of the upper limb
3. Ongoing use of central nervous system (CNS)-active medications
4. Ongoing use of psychoactive medications, such as stimulants, antidepressants, and anti-psychotic medications
5. Botox or phenol alcohol treatment within 12 weeks of enrollment
6. Pregnancy in women, as determined by self-report
7. History of spinal cord injury or weakness
8. Chronic pain
9. Peripheral neuropathy including insulin dependent diabetes as determined by case history
10. Presence of additional potential tsDCS risk factors:

    * Damaged skin at the site of stimulation (i.e., skin with ingrown hairs, acne, razor nicks, wounds that have not healed recent scar tissue, broken skin, etc.)
    * Presence of an electrically, magnetically or mechanically activated implant (including cardiac pacemaker), an intracerebral vascular clip, or any other electrically sensitive support system
    * Highly conductive metal in any part of the body, including metal injury to the eye (jewelry must be removed during stimulation)
    * Past history of seizures or unexplained spells of loss of consciousness during the previous 36 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-09; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Feinstein Institute for Medical Research, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahmed Z. Trans-spinal direct current stimulation alters muscle tone in mice with and without spinal cord injury with spasticity. J Neurosci. 2014 Jan 29;34(5):1701-9. doi: 10.1523/JNEUROSCI.4445-13.2014. PMID 24478352
- [Background] Ahmed Z. Trans-spinal direct current stimulation modifies spinal cord excitability through synaptic and axonal mechanisms. Physiol Rep. 2014 Sep 28;2(9):e12157. doi: 10.14814/phy2.12157. Print 2014 Sep 1. PMID 25263206
- [Background] Samaddar S, Vazquez K, Ponkia D, Toruno P, Sahbani K, Begum S, Abouelela A, Mekhael W, Ahmed Z. Transspinal direct current stimulation modulates migration and proliferation of adult newly born spinal cells in mice. J Appl Physiol (1985). 2017 Feb 1;122(2):339-353. doi: 10.1152/japplphysiol.00834.2016. Epub 2016 Dec 8. PMID 27932680
- [Background] Winkler T, Hering P, Straube A. Spinal DC stimulation in humans modulates post-activation depression of the H-reflex depending on current polarity. Clin Neurophysiol. 2010 Jun;121(6):957-61. doi: 10.1016/j.clinph.2010.01.014. Epub 2010 Feb 11. PMID 20153248
- [Background] Bocci T, Vannini B, Torzini A, Mazzatenta A, Vergari M, Cogiamanian F, Priori A, Sartucci F. Cathodal transcutaneous spinal direct current stimulation (tsDCS) improves motor unit recruitment in healthy subjects. Neurosci Lett. 2014 Aug 22;578:75-9. doi: 10.1016/j.neulet.2014.06.037. Epub 2014 Jun 23. PMID 24970753
- [Background] Truini A, Vergari M, Biasiotta A, La Cesa S, Gabriele M, Di Stefano G, Cambieri C, Cruccu G, Inghilleri M, Priori A. Transcutaneous spinal direct current stimulation inhibits nociceptive spinal pathway conduction and increases pain tolerance in humans. Eur J Pain. 2011 Nov;15(10):1023-7. doi: 10.1016/j.ejpain.2011.04.009. Epub 2011 May 14. PMID 21576030
- [Background] Cogiamanian F, Vergari M, Pulecchi F, Marceglia S, Priori A. Effect of spinal transcutaneous direct current stimulation on somatosensory evoked potentials in humans. Clin Neurophysiol. 2008 Nov;119(11):2636-40. doi: 10.1016/j.clinph.2008.07.249. Epub 2008 Sep 10. PMID 18786856
- [Derived] Paget-Blanc A, Chang JL, Saul M, Lin R, Ahmed Z, Volpe BT. Non-invasive treatment of patients with upper extremity spasticity following stroke using paired trans-spinal and peripheral direct current stimulation. Bioelectron Med. 2019 Jul 23;5:11. doi: 10.1186/s42234-019-0028-9. eCollection 2019. PMID 32232101

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants received both the anodal and sham trans-spinal direct current stimulation + peripheral direct current stimulation (tsDCS + pDCS) conditions, and sequence of stimulation conditions was the same across participants, with sham stimulation preceding active stimulation.
Groups:
- Sham Doublestim, Then Anodal Doublestim: Participants underwent 2-3 baseline evaluations, then received 5 daily, consecutive 20 min sessions of sham Doublestim (trans-spinal direct current stimulation + peripheral direct current stimulation). After a washout period of 1 week, sham FU measures were collected. Participants then received 5 daily, consecutive 20 min sessions of anodal Doublestim (trans-spinal direct current stimulation + peripheral direct current stimulation), and again underwent follow-up measures 1 week after the anodal intervention. For all participants, the sham condition preceded the anodal Doublestim condition.
Period: Baseline
Arm/Group | Sham Doublestim, Then Anodal Doublestim
Started | 26
Completed | 24 (Two participants (pts) dropped out after consent due to hospitalizations unrelated to the study.)
Not Completed | 2
Not completed — Adverse Event | 2
Period: Sham Doublestim (5days)
Arm/Group | Sham Doublestim, Then Anodal Doublestim
Started | 24
Completed | 24
Not Completed | 0
Period: Sham FU (7days)
Arm/Group | Sham Doublestim, Then Anodal Doublestim
Started | 24
Completed | 24
Not Completed | 0
Period: Anodal Doublestim (5 Days)
Arm/Group | Sham Doublestim, Then Anodal Doublestim
Started | 24
Completed | 23
Not Completed | 1
Not completed — Adverse Event | 1
Period: Anodal FU (7 Days)
Arm/Group | Sham Doublestim, Then Anodal Doublestim
Started | 23
Completed | 19
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Groups:
- Sham Doublestim, Then Anodal Doublestim: Crossover design study: Participants first received 5 daily, consecutive 20 min sessions of sham Doublestim (trans-spinal direct current stimulation + peripheral direct current stimulation). After a washout period of 1 week, they then received 5 daily, consecutive 20 min sessions of anodal Doublestim (trans-spinal direct current stimulation + peripheral direct current stimulation).
Arm/Group | Sham Doublestim, Then Anodal Doublestim
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 20
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline in Area Under the Curve for Objectively Measured Spastic Catch Response of the Wrist Flexors at Fast Speed
Description: Subjects' wrists were passively extended at fast speed by a stepper motor to induce a spastic catch response, and its resistance torque was calculated in Newton meters (Nm). Mean percent change from baseline in the area under the curve for the resistance torque were compared across two timepoints (final session at day 5 and 1 week follow-up) in two conditions (sham vs. anodal Doublestim)
Time Frame: baseline, final session at day 5, 1 week FU
Population: Three subjects (out of 19) were found to be significant outliers for normality testing, and were consequently removed from analysis.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Sham Doublestim | Anodal Doublestim
Number analyzed (Participants) | 16 | 16
percent change
  Mean percent change at final session (day 5) | 13.678 (5.537) | -8.783 (4.911)
  Mean percent change at 1 week follow-up (FU) | 15.927 (5.537) | -16.333 (6.180)
Statistical Analysis 1: Comparison: Sham Doublestim vs Anodal Doublestim; Test type: Equivalence — Statistical analysis for mean percent change from baseline in area under the curve for the resistance torque measure across 2 conditions (anodal vs. sham Doublestim) and at 2 timepoints (final session at day 5 and 1 week FU). Null hypothesis is that there was no difference in mean percent change in area under the curve between anodal and sham Doublestim conditions. A significance level of 0.05 was used (two-sided); p = 0.004, ANOVA — A 2x2 repeated measures ANOVA was performed with condition (mean percent change in anodal vs. sham condition) and time (final session at day 5 and 1 week FU in each condition) as factors. A significance level of 0.05 was used (two-sided)

2. Secondary Outcome: Mean Modified Tardieu Scale (MTS) Score
Description: The Modified Tardieu Scale (MTS) quantifies muscle spasticity for each joint at slow and fast velocities on a 0-5 point scale. MTS scores at fast velocity were summed across 11 joints of the upper extremity (for a total of 0-55 points), with lower scores indicating improved spasticity. Mean summed MTS scores (out of 55 total points) were compared across two timepoints (final session at day 5 and 1 week FU) in two conditions (sham vs. anodal Doublestim).
Time Frame: baseline, final session at day 5, 1 week FU
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Sham Doublestim | Anodal Doublestim
Number analyzed (Participants) | 16 | 16
scores on a scale
  mean score at final session (day 5) | 23.375 (0.275) | 21.625 (0.275)
  mean score at 1 week FU | 23.125 (0.275) | 21.975 (0.309)
Statistical Analysis 1: Comparison: Sham Doublestim vs Anodal Doublestim; Test type: Equivalence — Statistical analysis for mean Tardieu Scale Score summed across 11 joints of the upper extremity in 2 conditions (anodal vs. sham Doublestim) and at 2 timepoints (final session at day 5 and 1 week FU). Null hypothesis is that there was no difference in mean change between anodal and sham Doubleestim conditions. A significance level of 0.05 was used (two-sided); p = 0.003, ANOVA — A 2x2 repeated measures ANOVA was performed with condition (mean score in anodal vs. sham condition) and time (final session at day 5 and 1 week FU in each condition) as factors. A significance level of 0.05 was used (two-sided)

ADVERSE EVENTS:
Time Frame: eight weeks for each subject
Description: Safety population included all participants who enrolled in study.
Groups:
- Baseline: Prior to any treatment interventions, participants performed 2-3 clinical and objective measure baseline evaluations.
- Sham Doublestim (5 Days) + Sham FU (7days); Anodal Doublestim (5 Days) + Anodal FU (7days): Following baseline evaluations, participants first received 5 daily, consecutive 20 min sessions of sham Doublestim (trans-spinal direct current stimulation + peripheral direct current stimulation). After a washout period of 1 week, they received a sham follow-up (FU) measure 7 days post-sham stimulation. Participants then received 5 daily, consecutive 20 min sessions of anodal Doublestim (trans-spinal direct current stimulation + peripheral direct current stimulation), followed by an anodal FU measure 7 days post-anodal Doublestim.
Arm/Group | Baseline | Sham Doublestim (5 Days) + Sham FU (7days) | Anodal Doublestim (5 Days) + Anodal FU (7days)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/26 | 0/24 | 2/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24 | 1/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline (N=26) | Sham Doublestim (5 Days) + Sham FU (7days) (N=24) | Anodal Doublestim (5 Days) + Anodal FU (7days) (N=24)
hypotensive vasovagal event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — A hypotensive vasovagal event (fainting episode) that occurred during a baseline clinical evaluation prior to any treatment sessions. The subject was excluded from the study and the event was judged not related to the device.
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Subject experienced an unrelated fall and hip fracture at home prior to receiving any stimulus in the study (sham or active), resulting in hospitalization and exclusion from the study.
seizure (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) — 2 subjects experienced a seizure 3-4 days after the fifth (final) active stimulation session. Both events were reported and deemed unrelated to study intervention.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline (N=26) | Sham Doublestim (5 Days) + Sham FU (7days) (N=24) | Anodal Doublestim (5 Days) + Anodal FU (7days) (N=24)
persistent skin redness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Subject experienced moderate-severe neck redness immediately following stimulation, with persistent mild neck redness 24 later. Given the durability of her neck redness, the subject was excluded from the study by the PI.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT03080454/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT03080454/ICF_001.pdf